CLINICAL TRIAL: NCT06104735
Title: Optimizing Spinal Cord Associative Plasticity to Enhance Response to Hand Training in Cervical Spinal Cord Injury
Brief Title: Finding the Best Combination of Brain and Spinal Cord Stimulation With Hand Training After Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bronx VA Medical Center (U.S. Federal Agency)
Collaborators: Bronx Veterans Medical Research Foundation, Inc (Other); New York State Department of Health (Other Government)
Responsible Party: Principal Investigator, Noam Y. Harel, Principal Investigator, Bronx VA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1777667
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Spinal Cord Injuries
Keywords: neuromodulation; spinal cord stimulation; task-oriented exercise; transcranial magnetic stimulation
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Exercise; SREBP cleavage-activating protein

STUDY DESIGN:
Intervention Model Description: Each participant will undergo multiple conditions and verifications in an "n-of-1" design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All participants (Experimental): Each participant will undergo varying conditions in separate phases to determine optimal: Pairing interval; Frequency; Number of bouts, Inter-bout spacing, and the order of SCAP when given in conjunction with task-oriented hand exercise.
  Interventions: Procedure: Synaptic Pairing Interval; Procedure: Frequency; Procedure: Bouts; Procedure: Spacing; Procedure: Exercise; Procedure: SCAP plus Exercise

INTERVENTIONS:
Procedure: Synaptic Pairing Interval — Optimize interstimulus pairing between brain and spinal cord stimulation.
Procedure: Frequency — Compare 2 Hz continuous to intermittent theta burst frequency
Procedure: Bouts — Compare effects of 1, 2, or 4 bouts of SCAP
Procedure: Spacing — Compare 6 versus 12 minutes of rest in between bouts of SCAP
Procedure: Exercise — Task-oriented hand exercises
Procedure: SCAP plus Exercise — Compare interleaved versus serial bouts of SCAP and exercise.

SUMMARY:
While physical exercise remains the foundation for any rehabilitation therapy, the team seeks to improve the benefits of exercise by combining it with the concept of "Fire Together, Wire Together" - when brain stimulation is synchronized with spinal cord stimulation, nerve circuits in the spinal cord strengthen - a phenomenon termed "Spinal Cord Associative Plasticity", or SCAP.

This project will build on the team's promising preliminary findings. When one pulse of brain stimulation is synchronized with one pulse of cervical spinal stimulation, hand muscle responses are larger than with brain stimulation alone or unsynchronized stimulation. However, the team does not know the best ways to apply SCAP repetitively, especially in conjunction with exercise, to increase and extend improvements in clinical function. Do ideal intervention parameters vary across individuals, or do they need to be customized?

The team will take a systematic approach with people who have chronic cervical SCI to determine each person's best combination of SCAP with task-oriented hand exercise. Participants will undergo up to 53 intervention, verification, and follow-up sessions over a period of 6 to 10 months each. The team will measure clinical and physiological responses of hand and arm muscles to each intervention.

Regaining control over hand function represents the top priority for individuals with cervical SCI. Furthermore, this approach could be compatible with other future interventions, including medications and cell-based treatments.

DETAILED DESCRIPTION:
See above.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-85 years.
* Must have stable prescription medication for 30 days prior to screening
* Must be able to: abstain from alcohol, smoking and heavy caffeine consumption on the day of each experiment; abstain from recreational drugs for the entirety of the study; commit to study requirements (i.e., 53 visits); provide informed consent.
* Score of 1-4 (out of 5) on manual muscle testing of finger extension, finger flexion, or finger abduction in left or right hand.

Exclusion Criteria:

* Personal or extensive family history of seizures;
* Ventilator dependence or patent tracheostomy site;
* History of stroke, brain tumor, brain abscess, or multiple sclerosis;
* History of severe head trauma requiring neurosurgery;
* History of implanted brain/spine/nerve stimulators, aneurysm clips, ferromagnetic metallic implants in the head (except for inside mouth); cochlear implants; cardiac pacemaker/defibrillator; intracardiac lines; currently increased intracranial pressure; or other contraindications to brain or spine stimulation;
* Significant coronary artery or cardiac conduction disease; recent history of myocardial infarction and heart failure with an ejection fraction of less than 30% or with a New York Heart Association Functional Classification of Class III or IV;
* Recent history (within past 6 months) of recurrent autonomic dysreflexia, defined as a syndrome of sudden rise in systolic pressure greater than 20 mm Hg or diastolic pressure greater than 10 mm Hg, without rise in heart rate, accompanied by symptoms such as headache, facial flushing, sweating, nasal congestion, and blurry vision (this will be closely monitored during all screening and testing procedures);
* History of significant hearing problems;
* History of bipolar disorder;
* History of suicide attempt;
* Active psychosis;
* Recent history (>1 year) of chemical substance dependency or significant psychosocial disturbance;
* Heavy alcohol consumption (greater than equivalent of 5oz of liquor) within previous 48 hours;
* Open skin lesions over the face, neck, shoulders, or arms;
* Pregnancy; and
* Unsuitable for study participation as determined by study physician.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 12 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Amplitude of motor evoked potential at the target muscle. | Through study completion, up to 10 months
  The primary neurophysiological outcome will be corticospinal excitability measured at the target muscle. The target muscle will be determined during the first evaluation session, with preference for first dorsal interosseous (FDI), abductor pollicis brevis (APB), or extensor carpi radialis (ECR) muscles based on muscle excitability and consistency. TMS recruitment curves will be collected. The amplitude of target muscle responses to TMS and spinal cord stimulation will be compared after the various interventions.

SECONDARY OUTCOMES:
Pinch and grip strength | Through study completion, up to 10 months
  Maximal isometric pinch strength will be measured in key-pinch (lateral edge of the index finger and the thumb) and tip-to-tip (tips of first and third finger) configurations using a pinch dynamometer. Grip strength will be measured using a hand dynamometer. For each type of pinch or grip, three trials will be conducted by holding the dynamometer with maximal volitional force for 3-5 seconds, with at least 30 seconds or more between trials. The highest achieved value will be used for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Noam Y Harel, MD, PhD, Principal Investigator — JAMES J. PETERS VAMC
Locations (1):
- James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York, United States